CLINICAL TRIAL: NCT05769894
Title: Is There an Association Between Non-cardiac Inflammatory Conditions and Dynamic Changes in Platelet Priming & Reactivity? A Prospective Observational Single Centre Study
Brief Title: Platelet Reactivity in Non-cardiac Inflammation A Prospective Observational Single Centre Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHMCAR0622
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Response; Platelet Aggregation, Spontaneous
MeSH Terms: conditions — Platelet Aggregation, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — -Blood samples for inflammatory markers (CRP, IL-6, CD-40, TNF alpha)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Fracture neck of femur: Trauma and Orthopaedics wards and the Emergency department will be screened for new admissions with fractured neck of femur proven by X-ray on admission, thereby identifying 20 participants according to eligibility criteria.
  Suitable patients will be approached about the study and given an information sheet. Later, when they have had enough time to consider, they will be enrolled if they are happy to provide written informed consent.
  Blood samples will be taken on the ward on admission, 24, 48 and 72 hours from admission and at 1 month.
  Blood will be collected in 4 tubes on each occasion. (1 x2ml 3.2% sodium citrate vacutainer, 1 x 6ml lithium heparin vacutainer. 2 x 5ml SST tubes for Inflammatory markers.) A detailed description of this is laid out below.
  Interventions: Other: No intervention given
- Patients > 70 years age admitted with chest infection: The Emergency department, Acute Medical Unit and medical wards will be screened for eligible participants whose primary diagnosis is chest infection (Acute bronchitis or Pneumonia). Aiming to recruit 20 participants.
  Acute Bronchitis is a lower respiratory tract infection causing inflammation in the bronchial airways It is a clinical diagnosis characterised by a cough with no evidence of pneumonia. The chest X-ray can be normal.
  Pneumonia is an infection of the lung tissue in which the air sacs in the lungs become filled with microorganisms, fluid and inflammatory cells, affecting the function of the lungs. 39 Patients will be selected according to symptoms, clinical diagnosis +/- Chest X-ray findings (Pneumonia only).
  Interventions: Other: No intervention given
- Healthy volunteers following COVID booster: Aiming to recruit 20 participants due to have a COVID vaccine at Southampton General Hospital. We are aiming to recruit 20 healthy volunteers meeting the criteria as per study eligibility.
  Interventions: Other: No intervention given
- Patient admitted with AMI within 6 weeks of inflammatory condition: Screening will include patients admitted with Type 1 or Type 2 MI or myocardial injury, as defined by the 4th Universal Definition, if they are within 6 weeks of one of the inflammatory conditions listed above.40 Suitable patients will be approached about the study and given an information sheet.
  Interventions: Other: No intervention given
- AMI secondary to stent thrombosis: Eligible patients will have been admitted with definite stent thrombosis according to the Academic Research Consortium definition. 41 Stent thrombosis is a complete occlusion of the artery secondary to thrombus inside the stent. ARC (Academic research consortium) has identified stent thrombosis detected by angiography as Definite stent thrombosis (ST). They also categorised stent thrombosis as early (up to 30 days from deployment), or late (30 days to 12 months from deployment).
  Suitable patients will be approached about the study and given an information sheet.
  Interventions: Other: No intervention given

INTERVENTIONS:
Other: No intervention given — No intervention is planned. Blood samples will be taken at different stages.

SUMMARY:
Non-cardiac acute and chronic inflammatory conditions are associated with high risk of acute myocardial infarction.

Specifically, there are reports of high prevalence of AMI and cardiac death in chronic conditions such as Rheumatoid arthritis, chronic gum disease, psoriasis and Chronic airway disease. Furthermore, there are intriguing temporal links between acute non-cardiac conditions, including fractured neck of femur and admission for chest infection in the elderly and subsequent risk of AMI within the next few weeks. Finally, a more recent association has been reported between COVID vaccination and acute thrombotic events.

In Summary, a link between acute non-cardiac inflammatory conditions and subsequent AMI in a near term envelope is established, but unexplained, and circumstantial evidence so far suggests a possible mechanism in terms of dynamic alteration in platelet reactivity. It is this concept we wish to explore further in the proposed set of experiments.

Our experiments may provide some insight into a potential mechanism of such an association, which could have implications for future tailored therapeutic interventions.

We will recruit 5 groups of patients, consistent with the data produced previously and the literature regarding disease models of non-cardiac inflammations. Aiming to recruit 20 patients per group with 100 candidates in total. Groups including:

1. Fracture neck of femur.
2. Patients >70 years age admitted with chest infection.
3. Healthy volunteers receiving fourth COVID booster vaccine.
4. Patients admitted with AMI within 6 weeks of (fractured neck of femur, chest infection Rheumatoid arthritis flare up, exacerbation of psoriasis and exacerbation of inflammatory bowel disease).
5. AMI secondary to stent thrombosis.

Study will be undertaken within the Cardiothoracic unit at University Hospital Southampton, the sponsor will be UHS Research and Development Department, UHS.

DETAILED DESCRIPTION:
BACKGROUND

Inflammation and Platelets

Cardiovascular disease (CVD) is the leading cause of death worldwide. Specifically, acute myocardial infarction (AMI) and acute ischaemic stroke are common causes of morbidity and mortality and are responsible for substantial healthcare costs. Whilst the underlying pathophysiology of atherosclerosis is now better understood as a chronic inflammatory process, the exact precipitants for the acute inflammation responsible for the acute event are still not fully explained. It has become clear that platelets play a key role in the pathophysiology of both atheroma formation and acute thrombus formation in AMI and stroke. Specifically, platelet activation is an integral component of initiation and amplification of the local vascular inflammatory response in these conditions. It is for this reason that routine antiplatelet therapy represents a mainstay of treatment for patients with coronary atheroma and especially for those treated with intracoronary stents.

Evidence for inter- and intra-individual variability in response to antiplatelets: dynamic reactivity

However, previous work from our group and others indicates that the response of individuals to both aspirin and P2Y12 inhibitors is idiosyncratic, so that some individuals may be relatively resistant to aspirin as well as clopidogrel, prasugrel and ticagrelor. Specifically, we have previously shown that patients on P2Y12 inhibitors for coronary stents with high on treatment platelet reactivity have elevated risk of stent thrombosis , and that individual responses can be modified using tailored therapy. Furthermore, our group has previously shown that the response to both aspirin and P2Y12 inhibitors is dynamic. Thus, there is a rebound Adenosine Diphosphate (ADP) response after clopidogrel is withdrawn in patients with drug-eluting stents. With regard to aspirin responses, we have reported that the response to arachidonic acid stimulation is variable within individuals, has some interaction with P2Y12 inhibitors, and that there appears to be a cyclo-oxygenase-dependent and -independent pathway for AA-induced platelet activity. Our previous data also suggest that the most commonly used near patient VerifyNow platelet test overestimates the response of patients to clopidogrel.

The WEST Group: Novel Assessments of Platelet Priming & Reactivity- Biomarkers of Individual Thrombotic Risk?

The research group led by Dr West has developed novel techniques for using (a) droplet microfluidics to assess hyper-reactivity of isolated platelets and (b) apply advanced single-platelet RNA sequencing methods to define an RNA signature for priming. These techniques have been subject to initial validation and show great promise as candidate biomarkers for predicting individual susceptibility to platelet-mediated thrombotic events such as acute myocardial infarction (AMI). For full background and previous data see Appendix.

This methodology is therefore complementary to our Thromboelastography (TEG)based assessment of platelet reactivity phenotype variability: we can validate the candidacy of the West method as biomarkers of thrombotic risk in these experiments.

Justification for our research question

For many reasons, no attempt is made in routine clinical practice to measure either the specific response of individuals to their antiplatelet drugs or the status of a patient's platelet reactivity at any moment in time. The development of tests that allowed both of these measurements to be made routinely could plausibly facilitate personalised detection and modification of high risk of bleeding or thrombotic events. The dynamic nature of an individual's platelet reactivity, and the possible contribution to acute thrombotic events is the focus for this series of experiments. Whilst it is not yet clear how the acute plaque erosion or rupture that precipitates AMI is initiated, the link to an acute inflammatory episode is apparent. Furthermore, an association has been demonstrated, described in detail below, between a number of non-cardiac acute and chronic inflammatory conditions, and subsequent risk of AMI. Specifically, there are reports of high prevalence of AMI and cardiac death in chronic conditions such as rheumatoid disease, chronic gum disease, psoriasis, chronic airways disease. Furthermore, as described below, there are intriguing temporal links reported between acute non-cardiac conditions, including fractured neck of femur and admission for chest infection in the elderly, and subsequent risk of AMI within the next few weeks. Finally, a more recent association has been reported between COVID vaccination and acute thrombotic events.

It is plausible that the "non-cardiac" inflammatory condition and/or event is, in actual fact, part of a disease process that incorporates dynamic changes in the arterial vascular bed and platelet reactivity, thereby providing the substrate for acute MI.

.

THEORETICAL FRAMEWORK Non-cardiac Inflammatory Conditions and Acute MI: known associations.

CVD and chest infection:

The annual incidence of community-acquired pneumonia (CAP) is 0.5-1% in United Kingdom, 22-42% of which requires hospitalization. The mortality rate of hospitalised patients with CAP is 5-14%, with higher mortality rates among elderly patients older than 84 years old (>50%).

Community acquired pneumonia is associated with raised inflammatory markers including CRP (>21.9 mg/dl), Pro-calcitonin and IL-6 (>169 pg/ml), with higher levels predicting treatment failure and mortality.

Furthermore, raised inflammatory markers were detected (CRP, TNF-alpha) in patients with viral upper respiratory tract infections.

Acute respiratory tract infection is associated with increased risk of acute myocardial infarction. Specifically, the first 28 days following respiratory tract infection, carries higher risk of cardiovascular events. In a case series study of 53709 patients with first or recurrent myocardial infarction, significant rise in MI incidence was noticed following acute respiratory tract infection with the highest rates being 3 days post infection.

Of interest, high on Treatment Platelet Reactivity was detected in patients with viral upper respiratory tract infection.

Studies assessing the link between MI and respiratory tract infection were mostly based on assessing GP records and questionnaires (history taking). Measuring levels of inflammatory markers during episodes of respiratory tract infection leading to MI was not tested.

Fractured Neck of Femur:

Hip fracture in the elderly population represents a substantial clinical and financial burden on our healthcare system, with high rates of morbidity and mortality. The mortality rate is 9% at 30 days post hip fracture and 33% at 1 year. A common complication of hip fractures is perioperative myocardial infarction. In one study, a Troponin rise was detected in 35.5% of patients and non-ST elevation Myocardial Infarction (NSTEMI) was more common than ST Elevation Myocardial Infarction (STEMI) in this cohort of patients. (23 vs 7) A significant troponin rise is a strong predictor of mortality in this patient group: a level above 0.04 μg/l is linked with six-fold risk of death. Highest troponin rise was specifically detected in the fourth post-operative day in the mortality group, compared to no significant rise in the alive group, with overall 1 year mortality detected in 37% of patients associated with Peri-operative troponin rise. 27,28 The mechanism behind the increased rate of myocardial infarction is not clear from current literature, but the suspicion is that there is a link to systemic inflammation induced by the fracture. There are weak data that some such patients may be hyporesponders to clopidogrel.

Rheumatoid arthritis flare up:

Rheumatoid arthritis (RA) affects approximately 1% of the adult western population. It is considered an independent risk factor for ischemic heart disease, with increased mortality due to accelerated coronary artery atherosclerosis.For example, rheumatoid arthritis was associated with a 38% increased incidence of myocardial Infarction compared to the general population in one series. The well described inflammatory process inherent to RA flare up, and the link to enhanced platelet reactivity, has been shown in a small study. Specifically, increased platelet reactivity to ADP only was noted in rheumatoid active group.

Major vascular surgery:

The Southampton group has previously described dynamic variability in platelet reactivity using TEG. Specifically, using TEG AUC 15 to assess 40 participants undergoing elective major vascular surgery (MVS) on aspirin, The investigators described a reduction in AA- and ADP-induced clotting in association with the acute vascular inflammatory reaction to surgery, with rebound reactivity (i.e., higher than baseline) at 3 months post op. The dynamic nature of these changes in platelet reactivity lends circumstantial support to the concept that this could play a role in pathological ischaemic events in susceptible individuals.

COVID vaccine:

The coronavirus disease 19 (COVID-19) pandemic has caused over 5 million deaths across the globe since 2019. COVID-19 infection is associated in some cases with thrombocytopenia due to platelet consumption, Disseminated Intravascular Coagulopathy (DIC) and thrombotic microangiopathy.

COVID-19 vaccines were approved in late 2020, with 5 billion individuals vaccinated so far. Increasing data have shown rare links between vaccines and thrombotic complications including cerebral sinus thrombosis and myocardial infarction. This may be related to the well-established systemic inflammatory reaction induced by the vaccine. Vaccine-induced immune thrombosis and thrombocytopenia (VITT) was identified in a small group of vaccinated individuals. In the few cases of acute coronary syndrome (ACS) post COVID-19 vaccination a cause-effect relation was not definitively established.

In summary, a link between acute non-cardiac inflammatory conditions and subsequent AMI in a near term envelope is established, but unexplained, and circumstantial evidence so far suggests a possible mechanism in terms of dynamic alteration in platelet reactivity. It is this concept that we wish to explore further in the proposed set of experiments.

RESEARCH QUESTION/AIM(S)

This study aims to assess the association between non-cardiac inflammatory conditions involving a vascular inflammatory reaction and dynamic platelet reactivity as determined using TEG6s device and two novel techniques for using (a) droplet microfluidics to assess hyper-reactivity of isolated platelets and (b) apply advanced single-platelet RNA sequencing methods to define an RNA signature for priming.

If our hypothesis is proven, our study will have demonstrated an association between (a) the presence, and possibly extent of, a dynamic change in individual platelet reactivity and blood clotting and (b) the concurrent vascular inflammatory status in a variety of non-cardiac inflammatory conditions.

Summary of study design:

* Suitable candidates meeting the eligibility criteria for participation in the study will be identified and approached by our research team during their hospital stay or vaccination hub visit (for COVID booster candidates).
* A member of the research team will explain the aim of the study, benefits, risks, and burdens with the potential participant. Candidates will be given sufficient time to decide if they would like to participate in the study.
* A written informed consent will be explained and signed by the candidate.
* First blood sample will be taken following consent, with further blood samples at 24, 48, 72 hours then 1 week or 1 month later depending on the group.
* All blood samples will be analysed as follows (i) After 30 mins of sampling, for platelet reactivity testing using the TEG 6s device, (ii) Single platelet/microfluidics analysis and (iii) Further samples will be sent for inflammatory markers testing.
* Participation in the study and follow up will end after the final follow up visit when final blood samples are collected.
* Data will be pseudonymised and analysed before being submitted to a peer-review journal.

The investigators will recruit 5 groups of patients, consistent with the data produced previously and the literature regarding disease models of non-cardiac inflammation. Details of blood testing and general inclusion and exclusion are summarised below.

In all cases, blood sampling will be for both assessment of platelet reactivity using TEG6S and for blood inflammatory markers (CRP, IL6, TNF alpha and CD40)

1. Group 1: Fractured neck of femur (n=20). Trauma and Orthopaedics wards and the Emergency department will be screened for new admissions with fractured neck of femur proven by X-ray on admission, thereby identifying 20 participants according to eligibility criteria.

   Suitable patients will be approached about the study and given an information sheet. Later, when they have had enough time to consider, they will be enrolled if they are happy to provide written informed consent.

   Blood samples will be taken on the ward on admission, 24, 48 and 72 hours from admission and at 1 month.

   Blood will be collected in 4 tubes on each occasion. (1 x2ml 3.2% sodium citrate vacutainer, 1 x 6ml lithium heparin vacutainer. 2 x 5ml SST tubes for Inflammatory markers.) A detailed description of this is laid out below.
2. Group 2: Patients > 70 years age admitted with chest infection (n=20).

   The Emergency department, Acute Medical Unit and medical wards will be screened for eligible participants whose primary diagnosis is chest infection (Acute bronchitis or Pneumonia). Aiming to recruit 20 participants.

   Acute Bronchitis is a lower respiratory tract infection causing inflammation in the bronchial airways It is a clinical diagnosis characterised by a cough with no evidence of pneumonia. The chest X-ray can be normal.

   Pneumonia is an infection of the lung tissue in which the air sacs in the lungs become filled with microorganisms, fluid and inflammatory cells, affecting the function of the lungs. 39 Patients will be selected according to symptoms, clinical diagnosis +/- Chest X-ray findings (Pneumonia only).

   Suitable patients will be approached about the study and given an information sheet. Later, when they have had enough time to consider, they will be enrolled if they are happy to provide written informed consent.

   Blood samples will be taken on the ward on admission, 24, 48 and 72 hours from admission and at 1 month.

   Blood will be collected in 4 tubes on each occasion. (1 x 2ml 3.2% sodium citrate vacutainer, 1 x 6ml lithium heparin vacutainer. 2 x 5ml SST tubes for Inflammatory markers.) A detailed description of this is laid out below.
3. Group 3: Healthy volunteers receiving a COVID Booster vaccine. (n=20). Aiming to recruit 20 participants due to have a COVID vaccine at Southampton General Hospital. We are aiming to recruit 20 healthy volunteers meeting the criteria as per study eligibility. Information sheet will be given to participant and they will have sufficient time to consider participating or not in the study.

   Blood samples will be taken directly after injection of COVID booster dose. Participants will be invited to attend 24-, 48-, and 1-week post booster injection to our research office on Cath lab day unit for blood sampling.

   Blood will be collected in 4 tubes on each occasion. 1x 2ml 3.2% sodium citrate vacutainer, 1 x 6ml lithium heparin vacutainer. 2 x 5ml SST tubes for Inflammatory markers.
4. Group 4: Patients admitted with AMI within 6 weeks of:

   1. Fractured neck of femur
   2. Chest Infection
   3. Rheumatoid arthritis flare up
   4. Exacerbation of psoriasis
   5. Exacerbation of inflammatory bowel disease

   Screening will include patients admitted with Type 1 or Type 2 MI or myocardial injury, as defined by the 4th Universal Definition, if they are within 6 weeks of one of the inflammatory conditions listed above.40 Suitable patients will be approached about the study and given an information sheet. Later, when they have had enough time to consider, they will be enrolled if they are happy to provide written informed consent.

   Blood samples will be taken on the ward on admission, 24, 48 and 72 hours from admission and at 1 month.

   Blood will be collected in 4 tubes on each occasion. (1 x 2ml 3.2% sodium citrate vacutainer, 1 x 6ml lithium heparin vacutainer. 2 x 5ml SST tubes for Inflammatory markers.) A detailed description of this is laid out below.
5. Group 5: AMI secondary to stent thrombosis (n=20).

Eligible patients will have been admitted with definite stent thrombosis according to the Academic Research Consortium definition. 41 Stent thrombosis is a complete occlusion of the artery secondary to thrombus inside the stent. ARC (Academic research consortium) has identified stent thrombosis detected by angiography as Definite stent thrombosis (ST). They also categorised stent thrombosis as early (up to 30 days from deployment), or late (30 days to 12 months from deployment).

Suitable patients will be approached about the study and given an information sheet. Later, when they have had enough time to consider, they will be enrolled if they are happy to provide written informed consent.

Blood samples will be taken on the ward on admission, 24, 48 and 72 hours from admission and at 1 month.

Blood will be collected in 4 tubes on each occasion. (1 x 2ml 3.2% sodium citrate vacutainer, 1 x 6ml lithium heparin vacutainer. 2 x 5ml SST tubes for Inflammatory markers.) A detailed description of this is laid out below.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Indication for inclusion:

Group 1 fractured neck of femur Group 2 age >70yrs with chest infection Group 3 healthy volunteers receiving COVID booster dose Group 4 Acute myocardial infarction within 6 weeks from suffering (Fracture neck of femur, chest infection, rheumatoid arthritis flare-up, Psoriasis flare up or flare up of inflammatory bowel disease).

Group 5 Acute myocardial infarction secondary to stent thrombosis.

* Written Informed Consent to participate in the study.
* Antiplatelet Naïve on admission, except for Groups 4 & 5.

Exclusion Criteria:

* Surgery in an emergency setting.
* Liver failure. (From history and background, deranged Liver functions tests i.e AST/ALT)
* Renal failure requiring dialysis.
* Platelet count <150,000.
* Medications including steroids, anticoagulants, non-steroidal anti-inflammatory drugs, COX-inhibitors.
* Known malignancy.
* Pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Thorough explanation was described previously in identifying study population.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic platelet reactivity with non-cardiac inflammation | During the period of recruitment (Max 1 month for each patient)
  Detecting an association between dynamic platelet reactivity and vascular inflammatory status in a variety of non-cardiac inflammatory conditions

IPD SHARING:
Plan to Share IPD: Undecided